CLINICAL TRIAL: NCT02769520
Title: An Open-Label, Phase 2 Efficacy Study With Window of Opportunity Immune Assessment of Pembrolizumab in Relapsed, Locally Recurrent Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Efficacy Study of Pembrolizumab in Relapsed, Locally Recurrent Squamous Cell Cancer of the Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assuntina G. Sacco, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Assuntina G. Sacco, MD, Associate Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 151615
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: squamous cell carcinoma head and neck; pembrolizumab; cancer; SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg will be administered by IV infusion every 3 weeks up to 12 months or until disease progression
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg will be administered by IV infusion every 3 weeks up to 12 months or until disease progression
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to determine whether pembrolizumab, when given after salvage surgery, is effective in increasing the time a person with squamous cell cancer of the head and neck remains disease-free following locoregional disease recurrence.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether pembrolizumab, when given after salvage surgery, is effective in increasing the time a person with squamous cell cancer of the head and neck remains disease-free following locoregional disease recurrence.

This is a prospective, multi-center, open label, phase II study with a window of opportunity component in patients with recurrent squamous cell carcinoma of the head and neck (SCCHN) treated with adjuvant pembrolizumab following salvage surgery. Forty-five (45) patients will participate in this study to determine disease-free survival probability at 12 months. Secondary objectives include assessments of disease-free survival probability at 2 years, overall survival, adverse events and toxicity, and immune and molecular correlatives. For the window of opportunity component, patients will be randomized 3:1 in favor of receiving pembrolizumab 200 mg administered intravenously (IV) every three weeks for a maximum of two doses, versus placebo prior to salvage surgery. Approximately three to six weeks following the first dose of pembrolizumab, patients will undergo salvage surgery. Tumor tissue and blood will be collected at the time of surgery for immune correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Has pathologically confirmed SCCHN (oral cavity, oropharynx, larynx, hypopharynx) with evidence of local and/or locoregional recurrence. Laryngeal tumors will only be included if there is evidence of extralaryngeal spread, or there is associated nodal disease. For all other sites, superficial tumors can only be included if there is associated nodal disease.
* Has a documented disease-free interval (minimum 16 weeks) after initial curative intent therapy.
* Candidate for salvage resection.
* Able to provide tissue from diagnostic core biopsy of tumor lesion(s).
* Patient has adequate organ function.
* Female patient of childbearing potential has a negative serum or urine pregnancy within 72 hours prior to receiving the first dose of study medication.
* Female patient of childbearing potential agrees to use adequate birth control.
* Male patient with a partner of childbearing potential agrees to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Patient has disease of nasopharyngeal carcinoma histology.
* Patient has evidence of metastatic disease.
* Patient is currently receiving or has received another investigational agent within 4 weeks prior to study Day 1.
* Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
* Patient has a known history of active TB (Bacillus Tuberculosis).
* Patient has received a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or baseline) from adverse events due to a previously administered agents.
* Patient has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1.
* Patients who have had major surgery or have insufficient recovery from surgical-related trauma or wound healing within 14 days from study Day 1.
* Patient has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Patient has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Notes: (1) Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment within the past 2 years are not excluded. (2) Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patient has a known history of, or any evidence of active, non-infectious pneumonitis.
* Patient receives chronic steroid use > 10 mg prednisone (or steroid equivalent) daily.
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Patient has received immunotherapy with inhibitors of PD-1 or PD-L1, or CTLA-4 blocking antibodies within 4 months prior to study Day 1.
* Patient has known active Hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known Human Immunodeficiency Virus (HIV) carrier (HIV 1/2 antibodies).
* Patient has interstitial lung disease.
* Patient is an appropriate candidate for adjuvant radiation after salvage therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 12 months
  Disease-Free Survival

SECONDARY OUTCOMES:
Disease-Free Survival at 2 years | 2 years
  Disease-Free Survival at 2 years
Overall Survival | 3 years
  Overall Survival
Safety: Incidence of Adverse Events, Serious Adverse Events, and Treatment Delays | 3 years
  Safety: Incidence of Adverse Events, Serious Adverse Events, and Treatment Delays

CONTACTS AND LOCATIONS:
Overall Officials: Assuntina Sacco, MD, Study Director — University of California, San Diego
Locations (3):
- United States (3):
  - UCSD Moores Cancer Center, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - University of California Los Angeles, Torrance, California

IPD SHARING:
Plan to Share IPD: No